CLINICAL TRIAL: NCT06696508
Title: Comparison Between Classic Laparoscopic Dismembered Pyeloplasty and Insitu Spatulation with Pre-Dismembering Ureteropelvic Angle Suturing; a Prospective Controlled Randomized Study.
Brief Title: Comparison Between Classic Laparoscopic Dismembered Pyeloplasty and Insitu Spatulation with Pre-Dismembering Ureteropelvic Angle Suturing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelghany, lecturer, urology department ,faculty of medicine , cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-60-2024
Record Dates: First submitted 2024-09-20; First posted 2024-11-20 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Pyeloplasty; Ureteropelvic Junction Obstruction
Keywords: pyeloplasty, laparoscopic pyeloplasty ,; dismembered pyeloplasty; ureteropelvic junction obstruction
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insitu spatulation and pre-dismembering ureteropelvic angle suturing during laparoscopic pyeloplasty (Experimental): After proper dissection of the PUJ, the anterior wall of the renal pelvis was incised.
  The incision continued downwards and laterally towards the PUJ and the lateral aspect of the ureter.
  In cases where crossing vessels were present, the pelvis with the PUJ and the uppermost part of the ureter were properly dissected from these vessels. This gave a wide room for pulling the pelvis upwards and gentle retraction of the crossing vessels allowing incision of the anterior wall of the pelvis and starting the spatulation of the PUJ. Spatulation could then continue to the upper ureter behind the properly dissected and retracted vessels.
  After complete spatulation and before dismembering the PUJ, we made benefit of splinting the ureter in place; a Maryland grasper opened the lumen of the ureter and the first stitch was precisely placed from outside inwards at the proper angle of the ureteric spatulation using 5/0 Vicryl sutures.
  The posterior wall of the PUJ and the pelvis was then dismembered
  Interventions: Procedure: Insitu Spatulation with Pre-Dismembering Ureteropelvic Angle Suturing during laparoscopic pyeloplasty
- the classic approach group (Active Comparator): the PUJ was dismembered after proper dissection, the lateral aspect of the ureter was spatulated and the first stich was also placed in the spatulation angle from outside inwards. All these steps were done after the discontinuation of the ureter and the pelvis, losing the benefit of ureteric splinting and orientation
  Interventions: Procedure: Classic Laparoscopic Dismembered Pyeloplasty

INTERVENTIONS:
Procedure: Insitu Spatulation with Pre-Dismembering Ureteropelvic Angle Suturing during laparoscopic pyeloplasty — After proper dissection of the PUJ, the anterior wall of the renal pelvis was incised.
  The incision continued downwards and laterally towards the PUJ and the lateral aspect of the ureter.
  In cases where crossing vessels were present, the pelvis with the PUJ and the uppermost part of the ureter were properly dissected from these vessels. This gave a wide room for pulling the pelvis upwards and gentle retraction of the crossing vessels allowing incision of the anterior wall of the pelvis and starting the spatulation of the PUJ. Spatulation could then continue to the upper ureter behind the properly dissected and retracted vessels.
  After complete spatulation and before dismembering the PUJ, we made benefit of splinting the ureter in place; a Maryland grasper opened the lumen of the ureter and the first stitch was precisely placed from outside inwards at the proper angle of the ureteric spatulation using 5/0 Vicryl sutures.
  The posterior wall of the PUJ and the pelvis was then dismembered
  Arms: Insitu spatulation and pre-dismembering ureteropelvic angle suturing during laparoscopic pyeloplasty
Procedure: Classic Laparoscopic Dismembered Pyeloplasty — the PUJ was dismembered after proper dissection, the lateral aspect of the ureter was spatulated and the first stich was also placed in the spatulation angle from outside inwards. All these steps were done after the discontinuation of the ureter and the pelvis, losing the benefit of ureteric splinting and orientation
  Arms: the classic approach group

SUMMARY:
Background and Rationale One of the most challenging steps in laparoscopic pyeloplasty is the ureteral spatulation in addition to the apical suture placement. In this study we will describe a simplified technique to facilitate these tricky steps in order to avoid ureteral shortening, loss of orientation, to minimize ureteral manipulations and to avoid the early loss of pelvic tissue.

Objectives:

To describe our technique and assess its feasibility and its benefit to facilitate the ureteropelvic anastomosis in laparoscopic pyeloplasty.

Study population , Sample size :

Patients with UPJO indicated for laparoscopic pyeloplasty 50 patient

Study Design:

A Prospective Controlled Randomized Study.

patients and methods : children less than ten years old with significant primary UPJ obstruction who were candidates for laparoscopic pyeloplasty were prospectively enrolled in this study. PUJ obstruction was discovered either incidentally on abdominal imaging or due to clinical presentation and complaints of the patients. Pre operative imaging was done for all patients in the form of ultrasonography, CT urography (CTU) and renal isotope scanning using Technetium-99m Diethylene Triamine Penta Acetic acid (Tc-99m DTPA). The indication for intervention was based either clinically on the patients' complaints or due to radiological signs of significant obstruction necessitating repair. Those who presented clinically were complaining of significant loin pain or repeated urinary tract infections. As regards the radiological indications of intervention, significant obstruction was deemed in cases of high grade or increase of hydronephrosis affecting the parenchymal thickness or echogenicity in repeated ultrasonography, marked hydronephrosis with delayed secretion of the intravenously injected contrast in CTUT or split renal function affection with obstructed pattern (t½ >20 min with rising curve) in diuretic renal isotope scanning.

Patients with previous abdominal surgery, concomitant secondary calculi or anatomically abnormal kidneys (as ectopic or horseshoe kidneys) were excluded from the study.

The patients were randomized into one of two study groups: (Group A) for classic laparoscopic dismembered pyeloplasty and (Group B) for laparoscopic in situ dismembered pyeloplasty. Randomization was done using closed envelopes.

The presence of crossing vessels did not contraindicate in situ spatulation and cases with aberrant vessels crossing the UPJ were randomized in both groups.

All cases were done by the same laparoscopic surgeon in the pediatric urology department. Data was prospectively collected after the Institutional Review Board approval of the study protocol.

Written informed consents were obtained from the patients' care givers before surgical intervention.

Surgical Technique Under general anaesthesia, routine retrograde study and insertion of ureteric catheter just below the PUJ with a guide wire passing into the pelvis were done in both groups.

In all cases, pyeloplasty was done through transperitoneal approach in lateral decubitus position via three 5 mm ports.

In the classic approach:

In brief, the PUJ was dismembered after proper dissection, the lateral aspect of the ureter was spatulated and the first stich was also placed in the spatulation angle from outside inwards. All these steps were done after the discontinuation of the ureter and the pelvis, losing the benefit of ureteric splinting and orientation.

As regards the second group:

After proper dissection of the PUJ, the anterior wall of the renal pelvis was incised.

The incision continued downwards and laterally towards the PUJ and the lateral aspect of the ureter.

In cases where crossing vessels were present, the pelvis with the PUJ and the uppermost part of the ureter were properly dissected from these vessels. This gave a wide room for pulling the pelvis upwards and gentle retraction of the crossing vessels allowing incision of the anterior wall of the pelvis and starting the spatulation of the PUJ. Spatulation could then continue to the upper ureter behind the properly dissected and retracted vessels.

After complete spatulation and before dismembering the PUJ, we made benefit of splinting the ureter in place; a Maryland grasper opened the lumen of the ureter and the first stitch was precisely placed from outside inwards at the proper angle of the ureteric spatulation using 5/0 Vicryl sutures.

The posterior wall of the PUJ and the pelvis was then dismembered and proper trimming and reduction of the pelvis were done if needed.

The same stich was placed at the most dependent site at the inferior angle of the pelvis from inside outwards.

In both groups:

In cases with aberrant crossing vessels :

All patients will underwent laparoscopic pyeloplasty with Insitu spatulation and pre-dismembering ureteropelvic angle suturing technique . Total operative time, stenting time, blood loss are all estimated. Patients will be followed after 3-6 months

DETAILED DESCRIPTION:
Background and Rationale:

Since described by Schuessler et al in 1993, laparoscopic pyeloplasty has become a good minimally invasive alternative to open approach with almost equivalent functional outcomes, relatively lower morbidity index and more smooth convalescence. Although has become familiar, laparoscopic dismembered pyeloplasty is still a demanding procedure with a steep learning curve especially for beginners. Beside intracorporeal suturing and knot tying, the ureteral manipulations for proper spatulation and the precise placement of the angle sutures are time consuming and technically challenging steps if done after ureteropelvic dismembering. Splinting of the ureter and preservation of its alignment not only can facilitate such steps and preserve the ureteric orientation to avoid its twisting, rotation or downward retraction but also protects against traumatizing or de-vascularizing the ureteric tissues especially the supposed anastomotic edges.

On the other hand, non-dismembered techniques like Fenger and flap pyeloplasty were described and adopted by many surgeons being technically easier due to the preservation of the alignment and continuity of the ureter and the renal pelvis. However, these techniques have much lower success rates.

Herein, we present a step wise modified technique for dismembered pyeloplasty in which the ureteric continuity remains intact to ensure its splinting and alignment for proper spatulation and precise placement of anastomotic angle's suture before dismembering. We also compared the intra operative and post operative outcomes to the classic dismembered technique.

Patients and Methods children less than ten years old with significant primary UPJ obstruction who were candidates for laparoscopic pyeloplasty were prospectively enrolled in this study. PUJ obstruction was discovered either incidentally on abdominal imaging or due to clinical presentation and complaints of the patients. Pre operative imaging was done for all patients in the form of ultrasonography, CT urography (CTU) and renal isotope scanning using Technetium-99m Diethylene Triamine Penta Acetic acid (Tc-99m DTPA). The indication for intervention was based either clinically on the patients' complaints or due to radiological signs of significant obstruction necessitating repair. Those who presented clinically were complaining of significant loin pain or repeated urinary tract infections. As regards the radiological indications of intervention, significant obstruction was deemed in cases of high grade or increase of hydronephrosis affecting the parenchymal thickness or echogenicity in repeated ultrasonography, marked hydronephrosis with delayed secretion of the intravenously injected contrast in CTUT or split renal function affection with obstructed pattern (t½ >20 min with rising curve) in diuretic renal isotope scanning.

Patients with previous abdominal surgery, concomitant secondary calculi or anatomically abnormal kidneys (as ectopic or horseshoe kidneys) were excluded from the study.

The patients were randomized into one of two study groups: (Group A) for classic laparoscopic dismembered pyeloplasty and (Group B) for laparoscopic in situ dismembered pyeloplasty. Randomization was done using closed envelopes.

The presence of crossing vessels did not contraindicate in situ spatulation and cases with aberrant vessels crossing the UPJ were randomized in both groups.

All cases were done by the same laparoscopic surgeon in the pediatric urology department. Data was prospectively collected after the Institutional Review Board approval of the study protocol.

Written informed consents were obtained from the patients' care givers before surgical intervention.

Surgical Technique Under general anaesthesia, routine retrograde study and insertion of ureteric catheter just below the PUJ with a guide wire passing into the pelvis were done in both groups.

In all cases, pyeloplasty was done through transperitoneal approach in lateral decubitus position via three 5 mm ports.

In the classic approach:

In brief, the PUJ was dismembered after proper dissection, the lateral aspect of the ureter was spatulated and the first stich was also placed in the spatulation angle from outside inwards. All these steps were done after the discontinuation of the ureter and the pelvis, losing the benefit of ureteric splinting and orientation.

As regards the second group:

After proper dissection of the PUJ, the anterior wall of the renal pelvis was incised.

The incision continued downwards and laterally towards the PUJ and the lateral aspect of the ureter.

In cases where crossing vessels were present, the pelvis with the PUJ and the uppermost part of the ureter were properly dissected from these vessels. This gave a wide room for pulling the pelvis upwards and gentle retraction of the crossing vessels allowing incision of the anterior wall of the pelvis and starting the spatulation of the PUJ. Spatulation could then continue to the upper ureter behind the properly dissected and retracted vessels.

After complete spatulation and before dismembering the PUJ, we made benefit of splinting the ureter in place; a Maryland grasper opened the lumen of the ureter and the first stitch was precisely placed from outside inwards at the proper angle of the ureteric spatulation using 5/0 Vicryl sutures.

The posterior wall of the PUJ and the pelvis was then dismembered and proper trimming and reduction of the pelvis were done if needed.

The same stich was placed at the most dependent site at the inferior angle of the pelvis from inside outwards.

In both groups:

In cases with aberrant crossing vessels in both groups, the ureter was translocated and the anastomosis was done in front of the crossing vessels.

The pelvis was then completely dismembered and the previously placed suture was tied.

Posterior wall anastomosis started first till a previously marked site at the healthy mucosa below the stenotic segment of the PUJ.

The stenotic segment of the PUJ was not trimmed until the anastomosis is completed. This allowed making use of this stenotic segment for traction without grasping the healthy mucosa of the ureter.

After completing the posterior wall anastomosis, the ureteric catheter was removed and a DJ stent was inserted on the guide wire in an antegrade rail way manner. The anterior wall anastomosis was then done.

A drain was then left and the ports' sites were closed at the end of the procedure.

Follow up All patients were monitored post operatively in a regular ward for vital signs, drains and urine output. In case of nil output (<50 cc) for 48 hours, drains were removed and the patients were discharged with the urethral catheter to be removed in the next follow up visit after 1 week.

DJ stents were planned to be removed after 4 weeks in both groups. Follow up abdominal ultrasonography was done on 3-, 6- and 12-months post operatively and diuretic renograms were done after 6 months.

Operative success was deemed in case of symptoms' resolution, if were preoperatively present, in addition to radiological amelioration of the degree of hydronephrosis in ultrasonography and improvement of split renal functions as well as diuretic curves in the follow up renal scintigraphy.

All patients' demographics, intra operative details and post operative data were recorded and analysed. As regards postoperative complications, the Clavien Dindo classiﬁcation was used

ELIGIBILITY:
Inclusion Criteria:

* patients candidates for laparoscopic pyeloplasty aged from 3 to 60 years old.

Exclusion Criteria:

* Patients undergoing pyeloplasty other than dismembered type.
* Patients with a history of previous ipsilateral surgery
* Patients undergoing pyeloplasty other than dismembered type.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
operative and post operative complication rate | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No